CLINICAL TRIAL: NCT06194318
Title: Phase 1, Placebo-controlled, Randomized, Observer-blind, First-in-human Study of Bivalent RSV Prefusion F Protein Vaccines (SCB-1019/SCB-1019T) in Healthy Adults
Brief Title: First-in-human Safety and Immunogenicity Study of SCB-1019 and SCB-1019T in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-1019-001
Record Dates: First submitted 2023-11-17; First posted 2024-01-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Syncytial Virus Vaccination
Keywords: Respiratory Syncytial Virus vaccination
MeSH Terms: interventions — arexvy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- group 1 (SCB-1019 low dose with Alum; young adults) (Experimental): 4 young adults (18-59 years old) will receive SCB-1019 (Low Dose with Alum) at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019
- group 2 (Placebo; young adults) (Placebo Comparator): 2 young adults (18-59 years old) will receive Placebo at Day 1
  Interventions: Biological: placebo
- group 3 (SCB-1019 high dose with Alum; Young Adults) (Experimental): 4 young adults (18-59 years old) will receive SCB-1019 (high dose with Alum) at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019
- group 4 (Placebo; young adults) (Placebo Comparator): 2 young adults (18-59 years old) will receive Placebo at Day 1
  Interventions: Biological: placebo
- group 5 (SCB-1019 low dose without Alum; older adults) (Experimental): 10 older adults (60-85 years old) will receive SCB-1019 (low dose without Alum) at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019
- group 6 (SCB-1019 low dose with Alum; older adults) (Experimental): 10 older adults (60-85 years old) will receive SCB-1019 (low dose with Alum) at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019
- group 7 (Placebo; older adults) (Placebo Comparator): 4 older adults (60-85 years old) will receive Placebo at Day 1
  Interventions: Biological: placebo
- group 8 (SCB-1019 high dose without Alum; older adults) (Experimental): 10 older adults (60-85 years old) will receive SCB-1019 (high dose without Alum) at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019
- group 9 (SCB-1019 high dose with Alum; older adults) (Experimental): 10 older adults (60-85 years old) will receive SCB-1019 (high dose with Alum) at Day 1
  Interventions: Biological: Candidate vaccine, SCB-1019
- group 10 (Placebo; older adults) (Placebo Comparator): 4 older adults (60-85 years old) will receive Placebo at Day 1
  Interventions: Biological: placebo
- Group 11 (SCB-1019T high dose without Alum; older adults) (Experimental): 30 older adults (60-85 years old) will receive SCB-1019T (high dose without Alum) at Day
  Interventions: Biological: candidate vaccine, SCB-1019T
- Group 12 (AREXVY; older adults) (Active Comparator): 30 older adults (60-85 years old) will receive AREXVY at Day 1
  Interventions: Biological: AREXVY
- Group 13 (Placebo; older adults) (Placebo Comparator): 10 older adults (60-85 years old) will receive Placebo at Day 1
  Interventions: Biological: placebo
- Group 14 (SCB-1019T mid dose with Alum; older adults) (Experimental): 30 older adults (60-85 years old) will receive SCB-1019T (mid dose with Alum) at Day 1
  Interventions: Biological: candidate vaccine, SCB-1019T

INTERVENTIONS:
Biological: Candidate vaccine, SCB-1019 — The SCB-1019 vaccine contains RSV F protein subunits from the two dominant circulating strains, A strain (SCB-1019A) and B strain (SCB-1019B). SCB-1019A and SCB-1019B are recombinant RSV F-Trimer proteins engineered by fusing the ectodomain of RSV F protein with Trimer-Tag™
  Arms: group 1 (SCB-1019 low dose with Alum; young adults); group 3 (SCB-1019 high dose with Alum; Young Adults); group 5 (SCB-1019 low dose without Alum; older adults); group 6 (SCB-1019 low dose with Alum; older adults); group 8 (SCB-1019 high dose without Alum; older adults); group 9 (SCB-1019 high dose with Alum; older adults)
Biological: placebo — placebo
  Arms: Group 13 (Placebo; older adults); group 10 (Placebo; older adults); group 2 (Placebo; young adults); group 4 (Placebo; young adults); group 7 (Placebo; older adults)
Biological: candidate vaccine, SCB-1019T — The SCB-1019T vaccines contain RSV F protein subunits from the two dominant circulating strains, A and B strain. Antigens are recombinant RSV F-Trimer proteins engineered by fusing the ectodomain of RSV F protein with Trimer-Tag™
  Arms: Group 11 (SCB-1019T high dose without Alum; older adults); Group 14 (SCB-1019T mid dose with Alum; older adults)
Biological: AREXVY — AREXVY is a FDA-approved respiratory syncytial virus (RSV) vaccine for adults aged 60 and older. Developed by GSK, it targets the prefusion F glycoprotein to protect against lower respiratory tract disease caused by RSV.
  Arms: Group 12 (AREXVY; older adults)

SUMMARY:
First-in-human Safety and Immunogenicity Study of SCB-1019 and SCB-1019T in Healthy Adults

DETAILED DESCRIPTION:
A Phase 1, placebo-controlled, randomized, observer-blind, First-in-human Study to describe the Safety, reactogenicity and immunogenicity of a bivalent recombinant RSV vaccines (SCB-1019 and SCB-1019T) in healthy adults

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants 60 to 85 years of age at the screening visit.
2. Individuals willing and able to comply with study requirements, including all scheduled visits, vaccination, laboratory tests, and other study procedures.
3. Individuals willing and able to give an informed consent, prior to screening. Healthy participants as determined by medical history, physical examination, and clinical judgment of the investigator; participants with pre-existing stable medical conditions can be included.

Exclusion Criteria:

1. Acute disease or fever (≥38°C) at time of vaccination.
2. History of a severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccines.
3. Any progressive unstable or uncontrolled clinical conditions.
4. Any progressive or severe neurologic disorder, seizure disorder, or history of Guillain-Barré syndrome.

Please refer to Protocol for full list of Inclusion and Exclusion criteria.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the reactogenicity of SCB-1019, SCB-1019T compared with AREXVY vaccine | Within 7 days after vaccination
  Proportion of participants with local and systemic solicited AEs
Evaluate the safety tolerability of SCB-1019, SCB-1019T compared with AREXVY vaccine | Within 28 days after vaccination
  Proportion of participants with unsolicited AEs
Evaluate the safety and tolerability of SCB-1019, SCB-1019T compared with AREXVY vaccine | Throughout the study period, from enrollment to 6 months follow up
  Proportion of participants with SAEs, AESIs, MAAEs, AEs leading to early termination from the study
Evaluate the safety and tolerability of SCB-1019, SCB-1019T compared with AREXVY vaccine | Screening and Day 8
  Mean change and shift from baseline in hematology, biochemistry and coagulation parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Rook, MD, Principal Investigator — CMAX Clinical Research
Locations (2):
- Australia (2):
  - Fusion Clinical Research, Adelaide, Southern Australia
  - Linear Clinical Research, Nedlands, Western Australia